CLINICAL TRIAL: NCT01610388
Title: A Randomized, Double-Blind, Placebo-Controlled Repeat Dose Escalation, First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of Oral and Intravenous GSK1322322 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Oral and Intravenous GSK1322322 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 113376
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: healthy subjects; double-blind; FTIH; dose-escalation; absolute bioavailability; GSK1322322; BAL
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort A1 (Experimental): Single dose 60 minute infusion of 500mg IV GSK1322322/placebo followed by BID for 4 days
  Interventions: Drug: 500mg IV GSK1322322/placebo
- Cohort A2 (Experimental): Single dose 30 minute infusion of 500mg IV GSK1322322/placebo followed by BID for 4 days
  Interventions: Drug: 500mg IV GSK1322322/placebo
- Cohort B (Experimental): Initial single 1000mg oral GSK1322322/placebo dose, initial single dose 1000mg IV GSK1322322/placebo followed by BID for 4 days
  Interventions: Drug: 1000mg oral GSK1322322/placebo; Drug: 1000mg IV GSK1322322/placebo
- Cohort C (Experimental): Initial single 1500mg oral GSK1322322/placebo dose, initial single dose 1500mg IV GSK1322322/placebo followed by BID for 4 days
  Interventions: Drug: 1500mg oral GSK1322322/placebo dose; Drug: 1500mg IV GSK1322322/placebo
- Cohort D (Experimental): Single dose 2000mg IV GSK1322322J/placebo
  Interventions: Drug: 2000mg IV GSK1322322J/placebo
- Cohort E (Experimental): Single dose 3000mg IV GSK1322322J/placebo
  Interventions: Drug: 3000mg IV GSK1322322J/placebo
- Cohort F (Experimental): 1000mg IV GSK1322322J/placebo followed by BID for 4 days
  Interventions: Drug: 1000mg IV GSK1322322J/placebo

INTERVENTIONS:
Drug: 500mg IV GSK1322322/placebo — 500mg IV
  Arms: Cohort A1; Cohort A2
Drug: 1000mg oral GSK1322322/placebo — 1000mg oral
  Arms: Cohort B
Drug: 1000mg IV GSK1322322/placebo — 1000mg IV
  Arms: Cohort B
Drug: 1500mg oral GSK1322322/placebo dose — 1500mg oral
  Arms: Cohort C
Drug: 1500mg IV GSK1322322/placebo — 1500mg IV
  Arms: Cohort C
Drug: 2000mg IV GSK1322322J/placebo — 2000mg IV
  Arms: Cohort D
Drug: 3000mg IV GSK1322322J/placebo — 3000mg IV
  Arms: Cohort E
Drug: 1000mg IV GSK1322322J/placebo — 1000mg IV
  Arms: Cohort F

SUMMARY:
This first time in human (FTIH) study will be the first administration of GSK1322322 as an intravenous formulation and will investigate safety, tolerability, and pharmacokinetics in healthy subjects. One cohort of subjects will undergo bronchoalveolar lavage (BAL) for determination of GSK1322322 concentrations in lung with simultaneous comparison to plasma concentrations to evaluate drug penetration in the lung. The study will evaluate the absolute bioavailability of an oral tablet formulation as compared to the IV formulation.In addition, Amendment 01 will enable the investigation of an improved IV formulation (GSK1322322J mesylate salt) in an additional repeat dosing cohort and the supra-therapeutic cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included at the discretion of the Investigator only if the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the final follow up visit.
* Body weight greater than or equal to 50 kilograms and body mass index (BMI) between 18.5-29.9 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB less than 450 millisecond (msec); or QTcB less than 480 msec in subjects with Bundle Branch Block on Screening ECG

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Contraindications to bronchoalveolar lavage including hypercapnia greater than 50 mm Hg, refractory hypoxemia, reactive airway disease or asthma, unstable angina or acute myocardial infarction in the last 6 months, heart failure, and severe hemostatic alterations (Cohort C only).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, and within 5 days following discontinuation of GSK1322322 (for sensitive and narrow therapeutic index CYP3A4 substrates), unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Use of antacids, H2 blockers, proton pump inhibitors, vitamins, and iron supplements within 7 days prior to the first dose of study medication and for the duration of the trial, including follow-up.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to medications used in study, ie Atropine, Midazolam, Fentanyl, Lidocaine, Codeine (Cohort C only) that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters within a 56 day period.
* Pregnant females as determined by positive [serum or urine] test at screening or prior to dosing.

Lactating females.

* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate: males less than 45 and greater than 100 beats per minute (bpm) and females less than 50 and greater than 100bpm. PR interval less than 120 and greater than 220msec, QRS duration less than 70 and greater than 120 msec, and QTcB greater than 450msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (greater than or equal to 3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2012-01-26 (Actual); Study Completion 2012-01-26 (Actual)

PRIMARY OUTCOMES:
GSK1322322 safety parameters including the number of subjects with adverse events (AEs) | Cohort A up to 14 days; Cohort B and C up to 16 days
GSK1322322 safety parameters including absolute values and changes over time of clinical safety laboratory assessments. | Cohort A up to 14 days; Cohort B and C up to 16 days
GSK1322322 safety parameters including the change from baseline in vital signs (blood pressure (BP) and heart rate) | Cohort A up to 14 days; Cohort B and C up to 16 days
GSK1322322 safety parameters including change from baseline in electrocardiogram (ECG) parameters | Cohort A up to 14 days; Cohort B and C up to 16 days
GSK1322322 pharmacokinetic parameters (PK) after single oral dose, area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)). | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-∞)). | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose aximum observed concentration (Cmax). | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose time of occurrence of Cmax (tmax). | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose mean residence time (MRTpo) | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose apparent clearance after oral administration (CL/F) | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose apparent volume of distribution after oral administration (Vz/F) | Cohorts B and C on Day -2
GSK1322322 PK parameters after single oral dose terminal phase half-life (t 1/2). | cohort B and C on Day -2
GSK1322322 PK parameters after single IV dose area under the concentration-time curve from zero (pre-dose) to some fixed nominal time (12 hours) (AUC(0-12)). | Cohorts A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose area under the concentration-time curve from zero (pre-dose) to some fixed nominal time (24 hours) AUC(0-24) | Cohorts A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose AUC(0-t) | Cohorts A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose AUC(0-∞). | Cohorts A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose Cmax | Cohorts A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose mean residence time intravenous (MRTiv) | Cohort A, B, C, D, E on Day 1
GSK1322322 PK parameters after single IV dose t1/2 | Cohort A, B, C, D, E on Day 1
Absolute bioavailability will be determined by comparing oral AUC(0-∞) to IV AUC(0-∞) | Cohort B and C on Day -2 and Day 1
MAT of oral tablet will be determined (=MRTpo-MRTiv) | Cohort B and C on Day -2 and Day 1
After repeated IV doses, pharmacokinetic parameters including Area under the concentration-time curve over the dosing interval (AUC(0-τ)) | Cohorts A, B, C on Days 3 - 6
After repeated IV doses, pharmacokinetic parameters including Cmax | Cohorts A, B, C on Days 3 - 6
After repeated IV doses, pharmacokinetic parameters including CL | Cohorts A, B, C on Days 3 - 6
GSK1322322 concentrations in BAL obtained in epithelial lining fluid (ELF) and alveolar macrophages (AM) as compared to that in plasma | Cohort C Day 6

SECONDARY OUTCOMES:
GSK1322322 urine PK parameters: amount excreted (Ae) of unchanged GSK1322322, fraction of the dose excreted in the urine (fe) and renal clearance (CLr) following single dose IV administration from Period 2 and Period 3. | cohort B and C on Day 1 and 2
Day 6 GSK1322322 AUC(0-τ) compared to AUC(0-12) on Day 1 to evaluate the accumulation ratio following repeat IV administration of GSK1322322. | Cohorts A, B, C Day 6 and Day 1
Day 6 GSK1322322 AUC(0-τ) compared to AUC(0-∞) on Day 1 to evaluate time invariance following repeat IV administration of GSK1322322. | Cohorts A, B, C Day 6 and Day 1
GSK1322322 PK parameters: AUC(0-∞) on Day 1 and AUC(0-τ) on Day 6 following IV administration at different doses for the assessment of dose proportionality. | Cohorts A, B, C Day1 and 6
Microbiome analysis of stool prior to and after exposure to GSK1322322 | Cohort A, B,C, D, E single sample predose and single sample post dose
GSK1322322J safety parameters including the number of subjects with adverse events (AEs) | Cohort D and E up to 11 days, Cohort F up to 14 days
GSK1322322J safety parameters including absolute values and changes over time of clinical safety laboratory assessments | Cohort D and E up to 11 days; Cohort F up to 14 days
GSK1322322J safety parameters including the change from baseline in vital signs (blood pressure (BP) and heart rate) | Cohort D and E up to 11 days; Cohort F up to 14 days
GSK1322322J safety parameters including change from baseline in electrocardiogram (ECG) parameters | Cohort D and E up to 11 days: Cohort F up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Naderer OJ, Rodvold KA, Jones LS, Zhu JZ, Bowen CL, Chen L, Dumont E. Penetration of GSK1322322 into epithelial lining fluid and alveolar macrophages as determined by bronchoalveolar lavage. Antimicrob Agents Chemother. 2014;58(1):419-23. doi: 10.1128/AAC.01836-13. Epub 2013 Nov 4. PMID 24189245
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113376 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113376?search=study&study_ids=113376#rs
- Available data/document: Individual Participant Data Set: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register